CLINICAL TRIAL: NCT00417703
Title: A Prospective Investigation of the Intraocular Pressure Immediately Following Intravitreous Injection of Ranibizumab
Brief Title: Intraocular Pressure Immediately Following Intravitreous Injection of Ranibizumab
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Other Study IDs: 2006032
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Choroidal Neovascularization
Keywords: Intraocular Pressure; Intravitreous Injection; Ranibizumab
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will quantify the intraocular pressure elevation in the immediate time period following intravitreous injection. With more widespread use of intravitreous injections in patients that may require several injections per year, it is important to document the sudden increase in intraocular pressure, including the maximum intraocular pressure and the time required for the intraocular pressure to return to baseline. This data may be useful in stimulating additional studies to evaluate the long term ocular effects of repeated intravitreous injections.

We hypothesize that the intraocular pressure increases significantly following intravitreous injection and then returns to baseline during the initial thirty minutes following ranibizumab injection.

DETAILED DESCRIPTION:
We will assess the trend of intraocular pressure immediately following intravitreal injection of ranibizumab 0.5 mg (0.05 mL) by taking serial intraocular pressure readings every five minutes for thirty minutes after injection. This study is a prospective descriptive data collection consisting of measuring intraocular pressure immediately following intraocular injection, and at 5, 10, 15, 20, 25, and 30 minutes following injection of ranibizumab 0.5 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female Patients >18 years of age
2. Patients will have documented choroidal neovascular membranes on fluorescein angiogram and/or optical coherence tomography
3. Requiring treatment or maintenance therapy for choroidal neovascular membrane
4. Able and willing to provide written informed consent

Exclusion Criteria:

1. History of arterial occlusive disease of the eye.
2. History of advanced glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Westhouse, DO, Principal Investigator — Oklahoma State University Medical Center
Locations (1):
- Retina Support Services, Inc, Tulsa, Oklahoma, United States